CLINICAL TRIAL: NCT01459614
Title: Phase II Study of Gemcitabine/Taxotere/Xeloda (GTX) in Combination With Cisplatin in Subjects With Metastatic Pancreatic Cancer
Brief Title: Gemcitabine/Taxotere/Xeloda (GTX) With Cisplatin in Subjects With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Swim Across America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J11125; NA_00066595 (Other: JHM IRB); Swim Across America Laboratory (Other: Swim Across America)
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GTX-C (Experimental): Each cycle is 21 days (2 weeks Tx + 1 week off). Xeloda given days 1-14, Gemcitabine, Taxotere, and Cisplatin given days 4 and 11.
  For expansion cohort, each cycle is 28 days (2 weeks of Tx + 2 weeks off)
  Interventions: Drug: Gemcitabine; Drug: Taxotere; Drug: Xeloda; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — IV on Days 4 and 11
Drug: Taxotere — IV on Days 4 and 11
  Other Names: Docetaxel
Drug: Xeloda — orally, twice a day Days 1-14
  Other Names: Capecitabine
Drug: Cisplatin — IV Days 4 and 11
  Other Names: Platinol; CDDP

SUMMARY:
Primary Objectives

To assess the efficacy of the combination of gemcitabine, taxotere, and xeloda (GTX) with cisplatin in subjects with metastatic pancreatic cancer based on the progression-free survival (PFS) rate at 6 month.

Secondary Objectives

* To assess safety and characterize toxicities of the combination of GTX with cisplatin in subjects with metastatic pancreatic cancer.
* To estimate disease control rate (DCR), PFS, and overall survival (OS).
* To estimate a PFS rate of an expansion cohort testing an alternative schedule.

Study Design

This study is a single arm phase II study to assess the efficacy of GTX with cisplatin in subjects with metastatic pancreatic cancer. Approximately 38 evaluable subjects will be enrolled, 28 in the initial cohort and 10 in the expansion cohort

The study will have a safety run-in phase consisting of 6 subjects. To ensure that the combination is safe, the first six subjects will be treated at DL1 and observed for limiting toxicity for the first 2 cycles before continuation with further accrual. After the safety run-in, the study will be continuously monitored for adverse events.

The primary endpoint will be the PFS rate at 6 month, which is defined as the proportion of subjects alive, free of disease progression at 6 months. The treatment regimen would be considered of insufficient activity for further study in this population if PFS rate at 6 months is 50% or less, and the minimum required level of efficacy that would warrant further study with the proposed regimen is a 75% PFS rate at 6 months. The study design includes interim monitoring for futility using a predictive probability approach. We will stop the study early if given the information at the interim analysis, it is unlikely that the PFS rate at 6 months will be greater than 50% if the study continues to the end.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed metastatic pancreatic adenocarcinoma. Subjects with islet cell neoplasms are excluded. Subjects with mixed histology will be excluded.
* Subject has one or more tumors measurable by CT scan using RECIST 1.1 criteria. MRI is acceptable if a CT scan is contraindicated.
* Patient must be chemotherapy naïve or must have completed chemotherapy greater than 5 years prior to enrollment.
* Male or non-pregnant and non-lactating female of age >18 years
* ECOG performance status <1. ECOG 0 indicates that the patient is fully active and able to carry on all pre-disease activities without restriction; and, ECOG 1 indicates that the patient is restricted in physically strenuous activity but is ambulatory and able to carry out work of a light or sedentary nature
* Life expectancy of greater than 12 weeks.
* Subjects must have adequate organ and marrow function as defined below:

WBC ≥ 3,500/mcL Absolute Neutrophil Count ≥1,500/mcL Platelets ≥100 x 10^9/L Hemoglobin ≥ 9 g/d Total Bilirubin within normal institutional limits Alkaline phosphatase ≤ 2.5 x ULN (≤ 5 X ULN for subjects with documented liver metastases) AST(SGOT)/ALT(SGPT) ≤ 2.5 x ULN (≤ 5 X ULN for subjects with documented liver metastases) Creatinine within normal institutional limits OR Creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.

* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Willingness to undergo a tumor biopsy (implemented after the first 6 patients).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects who have had any prior chemotherapy within 5 years of enrollment
* Subjects who have had radiotherapy for pancreatic cancer.
* Age ≥ 76 years
* Subjects who are receiving or have received any other investigational agents within 28 days prior to Day 1 of treatment in this study.
* Subject has undergone major surgery, other than diagnostic surgery (i.e.--surgery done to obtain a biopsy for diagnosis or an aborted Whipple), within 28 days prior to Day 1 of treatment in this study.
* Subject has known brain metastases unless previously treated and well controlled for at least 3 months (defined as stable clinically, no edema, no steroids).
* History of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, taxotere, xeloda, or cisplatin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the subject to receive an experimental research drug.
* Subject has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Subject has a known history of infection with HIV, hepatitis B, or hepatitis C.
* Subject is pregnant or breast feeding.
* Subject is unwilling or unable to comply with study procedures.
* Subject with an unhealed surgical wound or other clinically significant wound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Wilbur HC, Durham JN, Lim SJ, Purtell K, Bever KM, Laheru DA, De Jesus-Acosta A, Azad NS, Wilt B, Diaz LA, Le DT, Wang H. Gemcitabine, Docetaxel, Capecitabine, Cisplatin, Irinotecan as First-line Treatment for Metastatic Pancreatic Cancer. Cancer Res Commun. 2023 Aug 28;3(8):1672-1677. doi: 10.1158/2767-9764.CRC-23-0230. eCollection 2023 Aug. PMID 37645623

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 patients were consented and screened. Of these, 5 were screen failures and 39 were eligible and assigned to receive treatment.
Groups:
- Primary Cohort (21 Day Cycle): Each cycle is 21 days. Xeloda (PO BID) given days 1-14, Gemcitabine (IV), Taxotere (IV), and Cisplatin (IV) given days 4 and 11.
- Expansion Cohort (28 Day Cycle): Each cycle is 28 days. Xeloda (PO BID) given days 1-14, Gemcitabine (IV), Taxotere (IV), and Cisplatin (IV) given days 4 and 11.
Period: Overall Study
Arm/Group | Primary Cohort (21 Day Cycle) | Expansion Cohort (28 Day Cycle)
Started | 29 | 10
Completed | 28 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Cohort (21 Day Cycle) | Expansion Cohort (28 Day Cycle) | Total
Number analyzed (Participants) | 29 | 10 | 39
Age, Continuous [Median (Full Range); unit: years] | 59 [43 to 75] | 67 [49 to 75] | 62 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 15
  Male | 16 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 8 | 36
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Disease Progression (Progression-Free Survival) at 6 Months
Description: PFS is defined as the percentage of patients with disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause at 6 months. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 6 months
Population: One patient was consented and enrolled, but was not considered evaluable per protocol, as he came off study prior to completing a cycle of treatment for reasons other than disease progression or death.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort (21 Day Cycle) | Expansion Cohort (28 Day Cycle)
Number analyzed (Participants) | 28 | 10
percentage of participants | 78.6 [59 to 92] | 30 [7 to 65]

2. Secondary Outcome: Number of Patients Experiencing a Grade 3 or Above Treatment-related Toxicity
Description: When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v4.03) will be counted only once for a given subject. AEs collected from time of first dose of study drug through 28 days after the last dose of study drug. The median duration of treatment was up to 23 months.
Time Frame: Up to 23 months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Cohort (21 Day Cycle) | Expansion Cohort (28 Day Cycle)
Number analyzed (Participants) | 29 | 10
Participants | 26 | 5

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of patients achieving a complete response (CR), partial response (PR), or stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: Up to 22 months
Population: Outcome was assessed for the Primary Cohort only per protocol. One patient was consented and enrolled, but was not considered evaluable per protocol, as he came off study prior to completing a cycle of treatment for reasons other than disease progression or death.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Primary Cohort (21 Day Cycle)
Number analyzed (Participants) | 28
Percentage of Participants | 89 [72 to 98]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the the number of months from the date of first dose to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause . Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: Up to 21 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Primary Cohort (21 Day Cycle) | Expansion Cohort (28 Day Cycle)
Number analyzed (Participants) | 28 | 10
Months | 8.4 [6.58 to 13.72] | 4.1 [3.74 to NA] — NA means that the upper bound confidence interval was not reached because the sample size was too small to estimate upper limit.

5. Secondary Outcome: Overall Survival (OS)
Description: OS (in months) will be measured from date of first dose until death (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: Up to 28 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Primary Cohort (21 Day Cycle)
Number analyzed (Participants) | 28
Months | 13.42 [10.48 to 20.13]

ADVERSE EVENTS:
Time Frame: AEs collected from time of first dose of study drug through 28 days after the last dose of study drug. The median duration of treatment was up to 23 months.
Description: AEs collected during protocol-specified visits, labs, and quality of life surveys.
Arm/Group | Primary Cohort (21 Day Cycle) | Expansion Cohort (28 Day Cycle)
All-Cause Mortality (participants affected / at risk) | 24/29 | 7/10
Serious Adverse Events (participants affected / at risk) | 5/29 | 1/10
Other Adverse Events (participants affected / at risk) | 29/29 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort (21 Day Cycle) (N=29) | Expansion Cohort (28 Day Cycle) (N=10)
febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
mucositis (Gastrointestinal disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0
neutrophil count decreased (Investigations) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 0
intracranial hemorrhage (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort (21 Day Cycle) (N=29) | Expansion Cohort (28 Day Cycle) (N=10)
Anemia (Blood and lymphatic system disorders) | 19 | 3
leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 10 | 3
Neutropenia (Blood and lymphatic system disorders) | 21 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 4
Ear pain (Ear and labyrinth disorders) | 2 | 0
Hearing impairment (Ear and labyrinth disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Blurred vision (Eye disorders) | 3 | 0
Vision Changes (Eye disorders) | 3 | 0
Watering eyes (Eye disorders) | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Anorexia (Gastrointestinal disorders) | 4 | 2
Bloating (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 15 | 7
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1
Hiccups (Gastrointestinal disorders) | 0 | 1
Indigestion or GERD (Gastrointestinal disorders) | 3 | 2
Mouth sores (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 16 | 3
Vomiting (Gastrointestinal disorders) | 10 | 6
Weight loss (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 0 | 1
Edema (General disorders) | 2 | 3
Fatigue (General disorders) | 12 | 2
Fever (General disorders) | 4 | 1
Infusion reaction (General disorders) | 0 | 1
Night sweats (General disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Thrush (Infections and infestations) | 3 | 4
ALT, increased (Investigations) | 3 | 0
AST, increased (Investigations) | 1 | 1
Bilirubin, increased (Investigations) | 0 | 1
Creatinine, increased (Investigations) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 16 | 4
Dizziness (Nervous system disorders) | 5 | 0
Dysgeusia (Nervous system disorders) | 17 | 3
Neuropathy (Nervous system disorders) | 12 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Smell Sensitivity (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 8
Blisters (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2
Nail Changes (Skin and subcutaneous tissue disorders) | 10 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes